CLINICAL TRIAL: NCT06677879
Title: A Prospective Cohort Study Comparing Proton and Photon Hypofractionated Radiotherapy for Left-sided Breast Cancer.
Brief Title: A Prospective Cohort Study of Proton and Photon Therapy for Left-sided Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, professor, Shanghai Proton and Heavy Ion Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-BCa2024-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; proton therapy; photon therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proton therapy (Experimental): Proton radiotherapy will be offered to patients who require adjuvant radiotherapy after lumpectomy or mastectomy for breast cancer.
  Interventions: Radiation: Proton radiotherapy
- photon therapy (Active Comparator): Photon radiotherapy will be offered to patients who require adjuvant radiotherapy after lumpectomy or mastectomy for breast cancer.
  Interventions: Radiation: Photon radiotherapy

INTERVENTIONS:
Radiation: Proton radiotherapy — Lumpectomy group: The total dose was 40.05Gy (RBE) , 2.67Gy (RBE) per fraction with 15 fractions. Once a day, five times a week. The tumor bed SIB to 48Gy (RBE).
  Mastectomy group: The total dose was 42.56Gy (RBE) , 2.66Gy (RBE) per fraction with 16 fractions. Once a day, five times a week.
  Arms: Proton therapy
Radiation: Photon radiotherapy — Lumpectomy group: The total dose was 40.05Gy, 2.67Gy per fraction with 15 fractions. Once a day, five times a week. The tumor bed SIB to 48Gy (RBE).
  Mastectomy group: The total dose was 42.56Gy, 2.66Gy per fraction with 16 fractions. Once a day, five times a week.
  Arms: photon therapy

SUMMARY:
The goal of this study is to investigate the differences in toxicity and efficacy between proton and photon hypofractionated radiotherapy following lumpectomy or mastectomy for breast cancer. The main questions it aims to answer are:

1. What is the difference in the incidence of radiation-related grade 2 or higher adverse events within two years following proton versus photon therapy after breast-conserving surgery?
2. What is the difference in the incidence of radiation-related grade 2 or higher adverse events within two years following proton versus photon therapy after mastectomy?

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer.
2. Indications for adjuvant radiotherapy following lumpectomy or mastectomy for left breast cancer:

   1. Post lumpectomy: Patients who have undergone lumpectomy with postoperative pathology staged as pT1-3 N1-3, excluding N3c.
   2. Post mastectomy: Patients who have undergone mastectomy, with postoperative pathology staged as pT1-3 N1-3, excluding N3c, and who have had an implant (prosthesis or tissue expander) placed.
3. Neoadjuvant therapy patients: Patients who have received neoadjuvant chemotherapy or endocrine/targeted therapy and have a postoperative stage of ypT1-3 N0-3, excluding N3c, requiring radiotherapy to the chest wall/breast and regional lymphatic drainage areas.
4. No distant metastasis.
5. Age range: 18-80 years.
6. Performance status: Eastern Cooperative Oncology Group (ECOG) score of 0-2.
7. Non-pregnant and non-lactating women.
8. Informed consent: Patients must provide written informed consent prior to receiving radiotherapy.

Exclusion Criteria:

1. Presence of Ductal Carcinoma In Situ (DCIS).
2. Tumor staging: Patients presenting with T4, N0, or N3c disease.
3. History of prior radiotherapy to the ipsilateral chest or breast.
4. Surgical margin status: Margins are either positive or close, defined as:

   Invasive carcinoma within 1 mm of the surgical margin.
5. Bilateral breast cancer: Patients with synchronous or previous contralateral breast cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The rate of patients who develop radiation-associated toxicity (≥ 2 degree) in 2 years | Until 2 years after radiotherapy
  We will record the incidence of ≥ 2 degree radiation-associated toxicity, such as breast or chest wall oedema, dermatitis, breast pain, esophagitis, rib fracture, radiation pneumonia and hypothyroidism and so on. The incidence of all the above is the primary outcome.

SECONDARY OUTCOMES:
Late toxicities after 2 years of radiotherapy | Until 5 years after radiotherapy
  Evaluation of long-term adverse effects (greater than 2 years) after radiotherapy (including radiation pulmonary fibrosis, radiation skin fibrosis, rib fracture, brachial plexus injury, upper limb lymphedema, heart injury, hypothyroidism, etc.)
Locoregional recurrence (LRR) | Until 5 years after treatment.
  To estimate and compare the rate of local recurrence between the proton and photon arms
Disease-free survival (DFS) | Until 5 years after treatment.
  Disease-free survival, defined as number of days from surgery until the first occurrence of local recurrence, distant metastases, tumor-related death, death without prior progression, or end of follow-up.
Overall survival (OS) | Until 5 years after treatment.
  Overall survival time, defined as number of days from date of initial diagnosis until death or end of follow-up.
uality of life, as measured by EORTC Quality of Life Questionnaires-B23 | During last week of radiotherapy, at 3 months post radiotherapy and 1,3 and 5 years post radiotherapy
  Impact on quality of life will be assessed by EORTC Quality of Life Questionnaires-B23；Which include functional domains, global health status and symptom scales.
Cosmetic outcome | Until 5 years after treatment.
  photographic cosmetic scores by BCCT.core

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China